CLINICAL TRIAL: NCT02521402
Title: Pilot Study to Evaluate Clinical Outcomes With the Use of Biovance, a Dehydrated Decellularized Human Amnion Membrane Allograft, Following Keloid Revision Surgery
Brief Title: Pilot Study to Evaluate Clinical Outcomes With the Use of Biovance Following Keloid Scar Revision Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Golla Center for Plastic Surgery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Golla-01-Keloid
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Keloid Scar
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Keloid Revision Surgery with Biovance (Other): All enrolled patients will have Biovance applied during Keloid Revision Surgery
  Interventions: Biological: Biovance

INTERVENTIONS:
Biological: Biovance — decellularized, dehydrated human amniotic membrane

SUMMARY:
The main purpose of this study is to see if there is clinical benefit of using Biovance in reduction of the recurrence of keloids when used to revise them. It will also assess the postoperative complications.

DETAILED DESCRIPTION:
To assess the performance of Biovance, patients will consulted regarding the history and previous treatment of their keloid. Once patients are deemed to be appropriate candidates, they will be enrolled in the study. Operatively, the old scar will be completely excised. Then the Biovance will be laid in the base of the wound. After this is performed, extensive undermining will be done to close the wound in layers.

All post-revision complications (including infection, incision dehiscence, hematoma, seroma, and wound necrosis) will be assessed and recorded by the investigator. Patients will be reviewed to obtain demographic and risk factor (such as age, body mass index, smoking) data. Data on adjuvant therapy use (previous surgeries, treatments for keloid scar) will be collected. Surgical technique details (such as incision size and closure technique) will also be recorded for each patient. Photographs documenting the pre-, intra- and post-revision clinical course of patients will be collected.

ELIGIBILITY:
Inclusion Criteria:

The subject has:

1. been diagnosed with a keloid scar
2. a keloid scar that is located on the face, neck, arm, trunk, or groin area
3. is between the ages of 21 and 80 years old
4. competency as an adult, per applicable state law who is willing to provide written informed consent
5. the intent and ability to return for all scheduled and required visits and follow recommended standard post surgical treatment for keloid scar excision.

Exclusion Criteria:

The subject has:

1. clinical evidence of infection of the keloid scar
2. any malignancy or a neoplasm at the keloid scar site
3. any significant comorbid disease that may interfere with wound healing, known active Hepatitis A, B, or C or Acquired Immune Deficiency Syndrome or is known to be infected with HIV, a known collagen disorder or autoimmune disease [including systemic lupus erythematosis (SLE), rheumatoid arthritis (RA),fibromyalgia, polymyositis, scleroderma, ankylosing spondylitis, dermatomyositis, osteogenesis imperfecta or the inherited disorders of Sjogren, Larsen, Raynaud, Ehlers-Danlos or Marfan syndrome]
4. received chemotherapy, radiotherapy, immunosuppressives or corticosteroids (greater than 10 mg prednisone-equivalent per day) within the past 30 days.
5. a known history of abuse of alcohol or drugs (prescribed or illegal), significant psychiatric personality or psychotic disorder requiring chronic psychotropic therapy, or gross noncompliance to recommended therapies
6. condition(s) that would adversely affect subject safety by following the protocol
7. any contraindication for use of Biovance

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of keloid scar recurrence after revision surgery with placement of Biovance | 1 year post-surgery
  Published data in the literature reporting on keloid scar incidence and recurrence without the use of Biovance may serve as a reference/historical control.

SECONDARY OUTCOMES:
Clinical outcomes of keloid scar revision surgery, including scar size and appearance | 1 year post-surgery
Incidence of complications (including infection, incision dehiscence, hematoma, seroma, and wound necrosis following revision surgery | 1 year post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dinakar Golla, MD, Principal Investigator — Golla Center for Plastic Surgery
Locations (1):
- Golla Center for Plastic Surgery, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Durani P, Bayat A. Levels of evidence for the treatment of keloid disease. J Plast Reconstr Aesthet Surg. 2008;61(1):4-17. doi: 10.1016/j.bjps.2007.05.007. Epub 2007 Jul 19. PMID 17644502
- [Result] Gauglitz GG, Korting HC, Pavicic T, Ruzicka T, Jeschke MG. Hypertrophic scarring and keloids: pathomechanisms and current and emerging treatment strategies. Mol Med. 2011 Jan-Feb;17(1-2):113-25. doi: 10.2119/molmed.2009.00153. Epub 2010 Oct 5. PMID 20927486
- [Result] Viera MH, Vivas AC, Berman B. Update on Keloid Management: Clinical and Basic Science Advances. Adv Wound Care (New Rochelle). 2012 Oct;1(5):200-206. doi: 10.1089/wound.2011.0313. PMID 24527306
- [Result] Alhady SM, Sivanantharajah K. Keloids in various races. A review of 175 cases. Plast Reconstr Surg. 1969 Dec;44(6):564-6. doi: 10.1097/00006534-196912000-00006. No abstract available. PMID 5352921
- [Result] Marneros AG, Norris JE, Watanabe S, Reichenberger E, Olsen BR. Genome scans provide evidence for keloid susceptibility loci on chromosomes 2q23 and 7p11. J Invest Dermatol. 2004 May;122(5):1126-32. doi: 10.1111/j.0022-202X.2004.22327.x. PMID 15140214
- [Result] Lee JY, Yang CC, Chao SC, Wong TW. Histopathological differential diagnosis of keloid and hypertrophic scar. Am J Dermatopathol. 2004 Oct;26(5):379-84. doi: 10.1097/00000372-200410000-00006. PMID 15365369
- [Result] Smiell JM, Treadwell T, Hahn HD, Hermans MH. Real-world Experience With a Decellularized Dehydrated Human Amniotic Membrane Allograft. Wounds. 2015 Jun;27(6):158-69. PMID 26061491